CLINICAL TRIAL: NCT04094389
Title: Comparison of Trigger Finger Orthotic Wearing Schedules: A Feasibility Study
Brief Title: Comparison of Trigger Finger Orthotic Wearing Schedules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, John Avery, OTR/L, CHT, Occupational Therapist, Certified Hand Therapist, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 1903804; IRB_00124056 (Other: University of Utah IRB)
Record Dates: First submitted 2019-09-15; First posted 2019-09-18 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: A randomized prospective pre-post test case series was chosen for this study. This case series will provide feasibility data in preparation for a randomized controlled study of this topic in the future.
  The primary research question for this case series is as follows: Do the three proposed orthotic wearing schedules provide varying results in the reduction of digital triggering severity and level of pain experienced by those with trigger finger? The following three orthotic wearing schedules will be investigated: only during waking hours, only while sleeping, and continuously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orthotic continuous wear group (Experimental): Participants in the continuous wear group will be instructed to wear their orthotic continuously around the clock as tolerated with removal for hygiene and home exercise program (HEP) performance.
  Interventions: Other: Orthotic continuous wear group
- Orthotic wear during waking hours only group (Experimental): Participants in the waking hours only group will be instructed to wear their orthotic during all waking hours as tolerated, with removal for hygiene, HEP performance, but not at night while sleeping.
  Interventions: Other: Orthotic wear during waking hours only group
- Orthotic wear only while sleeping group (Experimental): In the night-wear group, participants will be told to wear their orthosis only at night.
  Interventions: Other: Orthotic wear only while sleeping group

INTERVENTIONS:
Other: Orthotic continuous wear group — Performed exclusively for research purposes, participants will be assigned at entrance to the study to either wear the orthotic continuously, only during waking hours, or only while sleeping. There will be three participants in each of the three groups.
  Participants in the continuous wear group will be instructed to wear their orthotic continuously around the clock as tolerated with removal for hygiene and home exercise program (HEP) performance. Consistent with standard of care for the treatment of trigger finger with an orthotic, all nine of the participants will be instructed to wear their orthotic for at least six weeks, as tolerated, with continuation of orthotic wear up to 10 weeks if their triggering has not completely abated.
  Arms: Orthotic continuous wear group
Other: Orthotic wear during waking hours only group — Performed exclusively for research purposes, participants will be assigned at entrance to the study to either wear the orthotic continuously, only during waking hours, or only while sleeping. There will be three participants in each of the three groups.
  Participants in the waking hours only group will be instructed to wear their orthotic during all waking hours as tolerated, with removal for hygiene, HEP performance, but not at night while sleeping. Consistent with standard of care for the treatment of trigger finger with an orthotic, all nine of the participants will be instructed to wear their orthotic for at least six weeks, as tolerated, with continuation of orthotic wear up to 10 weeks if their triggering has not completely abated.
  Arms: Orthotic wear during waking hours only group
Other: Orthotic wear only while sleeping group — Performed exclusively for research purposes, participants will be assigned at entrance to the study to either wear the orthotic continuously, only during waking hours, or only while sleeping. There will be three participants in each of the three groups.
  In the night-wear group, participants will be told to wear their orthosis only at night. Consistent with standard of care for the treatment of trigger finger with an orthotic, all nine of the participants will be instructed to wear their orthotic for at least six weeks, as tolerated, with continuation of orthotic wear up to 10 weeks if their triggering has not completely abated
  Arms: Orthotic wear only while sleeping group

SUMMARY:
A randomized prospective pre-post test case series was chosen for this study. This case series will provide feasibility data in preparation for a randomized controlled study of this topic in the future.

The primary research question for this case series is as follows: Do the three proposed orthotic wearing schedules provide varying results in the reduction of digital triggering severity and level of pain experienced by those with trigger finger? The following three orthotic wearing schedules will be investigated: only during waking hours, only while sleeping, and continuously.

To examine the feasibility of the study the following questions are posed:

What was the length of time required to recruit nine eligible participants for the case series through the outpatient clinic utilized for this feasibility study? Based upon the rate of recruitment for the feasibility study, were the initial methods of recruitment adequate or did additional strategies need to be implemented to recruit a sufficient number of participants within the desired time frame? Were the orthotics utilized for the study comfortable to wear and functional for the participants while performing their activities of daily living? Were the number and type of adverse events including redness, edema, tingling, or numbness associated with orthotic wear similar across the groups, limited, non-serious, and did not interfere with orthotic wearing? Did participants wear their orthotics for the prescribed wearing schedule?

DETAILED DESCRIPTION:
Participants:

Nine participants will be recruited through a convenience sampling of patients as they become available through referral by physicians, physician assistants, and nurse practioners to the researcher's clinic for hand therapy, meet the study's eligibility criteria and provide informed consent to participate in the study. Medical records review will be performed by the principal investigator who will also be the potential participants' treating therapist.

At the onset of the study and as new referral sources become available, until all nine participants required for the study are enrolled, project flyers will be provided to referring physicians, physician assistants and nurse practioners for posting in their offices and providing to interested potential participants as desired.

Number of participants to be included and/or enrolled in this entire study, across all study locations: 20 Nine participants are needed for data analysis, however, 20 participants have been indicated for enrollment to cover for anticipated participant withdrawals and those who are lost to follow-up.

Age of Subjects: 18 to 85+ Vulnerable participant groups included: None Gender of Subjects: There are no gender-based enrollment restrictions for this study. Within the limitations imposed by the population of people with trigger finger, it is intended that there will be an equal gender distribution of the subjects included in the study.

Racial and Ethnic Origin: There are no race or ethnic-based enrollment restrictions for this study. Within the limitations imposed by the population of the study site, it is intended that this study will include sufficient enrollment of persons of diverse racial/ethnic backgrounds to ensure equitable selection

Study Design:

To examine the feasibility of the study the following questions are posed:

1. What was the length of time required to recruit nine eligible participants for the case series through the outpatient clinic utilized for this feasibility study?
2. Based upon the rate of recruitment for the feasibility study, were the initial methods of recruitment adequate or did additional strategies need to be implemented to recruit a sufficient number of participants within the desired time frame?
3. Were the orthotics utilized for the study comfortable to wear and functional for the participants while performing their activities of daily living?
4. Were the number and type of adverse events including redness, edema, tingling, or numbness associated with orthotic wear similar across the groups, limited, non-serious, and did not interfere with orthotic wearing?
5. Did participants wear their orthotics for the prescribed wearing schedule?

Procedures and Study Visits:

All procedures performed exclusively for the purposes of this study are performed in addition to the standard of care activities that would occur for all patients being provided with hand therapy for the treatment of a triggering upper extremity digit regardless of their participation in a study. These standard of care activities include standard clinical assessments, provision of an orthotic and wearing schedule, provision of a home exercise program and follow-up therapy sessions.

At the initial evaluation, consistent with standard of care activities that would occur for all patients regardless of their participation in a study, demographic data collected on each participant will include their age, gender, vocation, affected finger(s) and hand(s), duration of trigger finger symptoms, hand dominance, relevant co-existing diagnoses, and utilization of anti-inflammatory medications. Also consistent with standard of care procedures, the participants will be assessed on the outcome measures of severity of digital triggering and pain level during triggering at the initial evaluation to obtain a baseline and then reassessed weekly until their time of discharge to permit an assessment of the rate of recovery across time for each individual as well as for each of the three wearing schedules. If triggering is not evident (Froimson's [1999] grade I) or if the digit is unable to be actively unlocked (Froimson's [1999] grade III), the participants pain level during active composite digital flexion and extension through their full available active range of motion will be measured as per standard of care procedures. See table 1 for Froimson's (1999) grading of digital triggering severity.

During the initial evaluation, if the potential participant meets the study criteria they will be invited to participate in the study. If the potential participant agrees to participate in the study, they will then be provided with care that is unique to the study participants and needs to be performed at the time of the initial evaluation including the following: signing the consent will occur first, followed by completing the QuickDASH (Disabilities of the Arm, Shoulder and Hand Outcome Measure) being provided with an orthotic wearing schedule (which may be different if they do not agree to participate in the study), a home exercise program log and an orthotic wearing log.

All of the participant's questions relevant to the study and necessary to facilitate rational and thoughtful decision making by the participant will be answered prior to signing the consent form. Prior to obtaining consent, the prospective participants will be asked if they sufficiently understand the information provided in order to make an informed decision regarding whether or not to participate in the research.

Only for the purposes of this research study, the QuickDASH will be completed by the participant during their initial evaluation and then again during their discharge re-evaluation to permit a pre-intervention to post-intervention assessment.

As a standard of care activity that would normally occur for all patients with a triggering upper extremity digit regardless of their participation in a study, during the initial evaluation visit the participant will also be provided with a custom fabricated thermoplastic digital joint blocking orthosis. When the triggering of an index, middle ring or small digit is able to be immediately relieved by blocking the MCP joint into approximately 15 degrees of flexion, the participant will be provided with a custom MCP joint blocking orthotic that is secured to the proximal phalanx of the affected digit, crossing the MCP joint and blocking it at approximately 15 degrees of flexion and leaving the IP joints free. The number of MCP joints blocked will be determined by the number of triggering digits (Photos 1 and 4). If blocking of the affected index, middle, ring or small digit MCP joint does not relieve the triggering or if the participant is unable to tolerate wearing of the MCP blocking orthotic and the triggering is able to be relieved with isolated blocking of the PIP joint, the participant will be provided with a custom PIP joint blocking orthotic with the DIP and MCP joints left free (Photo 5). When the thumb is triggering and is able to be relieved of triggering by blocking the MCP joint into approximately 15 degrees of flexion, the participant will be provided with a custom MCP joint blocking with the IP and 1st carpometacarpal joint left free (Photo 7). If blocking of the thumb MCP joint alone does not relieve the triggering, both the MCP and IP joints will be blocked by the orthotic, with a sufficient amount of IP joint flexion permitted to allow thumb opposition to the index, middle, ring and small digits (Photo 8). If the participant is unable to tolerate wearing of the thumb MCP and IP blocking orthotic and triggering of the thumb is able to be relieved with blocking of the thumb IP joint alone, the participant will be provided with a thumb IP joint blocking orthotic (Photo 6). Figure 1 provides a flow chart illustrating the protocol that will be followed for this study to guide the decision-making process for selection of the most appropriate orthotic for the treatment of index through small finger triggering. Figure 2 provides a flow chart illustrating the protocol that will be followed for selecting an orthotic for the treatment of triggering thumbs.

Performed exclusively for research purposes, participants will be assigned at entrance to the study to either wear the orthotic continuously, only during waking hours, or only while sleeping. There will be three participants in each of the three groups. The first three participants will each be assigned to a different group through randomization. The remaining six participants will be assigned to one of the three groups based upon their Froimson's (1999) grade. The mean Froimson's (1999) trigger finger severity grade will be calculated for each group and participant assignments will be made as required to keep these means as equal as possible. Nine participants are needed for data analysis, however, 20 participants have been indicated for enrollment to cover for anticipated participant withdrawals and those who are lost to follow-up.

Participants in the continuous wear group will be instructed to wear their orthotic continuously around the clock as tolerated with removal for hygiene and home exercise program (HEP) performance. Participants in the day-wear group will be instructed to wear their orthotic during all waking hours as tolerated, with removal for hygiene, HEP performance, but not at night while sleeping. In the night-wear group, participants will be told to wear their orthosis only at night. Consistent with standard of care for the treatment of trigger finger with an orthotic, all nine of the participants will be instructed to wear their orthotic for at least six weeks, as tolerated, with continuation of orthotic wear up to 10 weeks if their triggering has not completely abated.

As a standard of care activity that would normally occur for all patients provided with an orthotic for the treatment of a triggering upper extremity digit regardless of their participation in a study, all participants will be educated on how to wear and care for the orthotic care and to discontinue wear of the orthotic and notify the principle investigator if they develop any adverse reactions including tingling, numbness, pain, edema or redness at orthotic wear site that lasts longer than 20 minutes. All participants will be provided with oral and written orthotic instructions that include their wearing schedule, precautions and care.

Performed for the purposes this study, to facilitate monitoring and measuring of orthotic wearing time, reasons for deviation from the wearing instructions and comfort of the orthotic, the participants will be instructed to keep a daily log of their orthotic donning and doffing consisting of time, date, reason for removing, comfort with wear, and functionality of the orthotic while performing their activities of daily living (Tarbhai et al., 2012; Valdes, 2012). The comfort of the orthotic will be rated on the following 0-3 scale: 0 (comfortable); 1 (uncomfortable with some activities); 2 (uncomfortable with most activities); 3 (uncomfortable with all activities). Adverse events including pain, redness, edema, tingling and numbness associated with wearing of the orthotic will be recorded on the daily log at the participants' earliest opportunity to increase the accuracy of the recording. Pain associated with wearing of the orthotic will be measured with the use of the NPRS. The participants functional use of their hand while wearing their orthotic to perform activities will be measured on a 0-3 scale: 0 (no difficulty); 1 (difficulty with some activities); 2 (difficulty with most activities); 3 (unable to do any activities while the orthotic is worn).

Participants will be instructed to complete the orthotic daily log at the following times: (a) The daily wear group as well as the continuous wear group will complete the log before retiring for the days longest sleeping period; (b) the participants wearing the orthotic only while sleeping will be instructed to fill out the log upon awakening. The orthotic daily log data will be collected by the investigator at six, eight and ten weeks after the participants' initial evaluation.

Consistent with standard of care activities, each participant will be provided with a HEP. Each HEP will include digital range of motion (ROM) and tendon gliding, including passive isolated and composite MCP, PIP and DIP flexion and extension, and active hook fist followed by active composite MCP and IP extension exercises (Colbourn et al., 2008; Evans et al., 1988; Valdes, 2012). If triggering is experienced during the HEP with the assigned active or passive ROM exercises, the participant will be instructed to only range the triggering digit through the active and / or passive non-triggering range.

Performed for the purposes of this study, to permit an estimation of the participants' compliance with their prescribed HEP performance schedule, the participants will be asked to complete a daily check-box log indicating their performance as most closely resembling one of the following: (a) as prescribed; (b) yes, but less than prescribed; or (c) not performed. The participants will be instructed to complete the HEP log before retiring for the days longest sleeping period. The HEP performance data will be collected by the investigator at six, eight and ten weeks after the participants' initial evaluation.

Follow-up therapy sessions, consistent with standard of care activities that would occur for all patients with a triggering upper extremity digit regardless of their participation in a study, will include the following: digital tendon gliding, ROM, edema reduction, HEP training and reinforcement as needed, inspection of the participant's skin for signs of adverse reaction to wearing of the orthotic, and modification of the orthotic or wearing schedule if necessary.

Procedure Frequency, Duration and Setting:

Participants will be provided with treatment sessions lasting approximately 45 minutes, occurring approximately twice per week, and for a duration of approximately 6-10 weeks with the end point of therapy being dependent upon complete resolution or plateauing of the participants progress with digital triggering. All study visits are also standard of care in that no subject in this study will require more visits than they would have required if they were not enrolled in this study.

The research procedures will be conducted at the Sharp Chula Vista Medical Center outpatient rehabilitation facility located at 752 Medical Center Court, Suite 303, Chula Vista, California, 91911.

Table 1: Froimson's (1999) grading of digital triggering severity Grade I - Pain associated with pre-triggering. Tenderness to palpation over the first annular pulley. Reported history of digital triggering, although not reproducible during clinical examination.

Grade II - Digital triggering occurs, although, digit can be unlocked with active extension.

Grade III - Digital triggering occurs and passive extension is necessary to unlock the digit, or active flexion is unable to be performed at the digit.

Grade IV - Digital triggering of the interphalangeal joint is unable to be unlocked with active or passive movement.

Data Analysis:

To assist with determining the feasibility of the study, the following data analyses will be reported through descriptive statistics:

The rate at which participants become available for the study. The participants' functional use of their hand and comfort while wearing their orthotic.

The participants' percentage compliance with their prescribed wearing schedules.

The participants' percentage compliance with their HEP performance schedule

Descriptive statistics will be utilized in this case series to describe the characteristics of participants' demographics, the adherence to the HEP, examine the data for changes in the outcome measurements for each of the participants across the 6 - 10 weeks of study, and to summarize the data to address the studies research question. The participants' pain and severity of digital triggering measurements, performed weekly across the 10 weeks of the study, will be calculated and reported for the mean and rate of change at each measurement period across time for each individual as well as for each of the three wearing schedule groups. The effect size for each group and between pairs of groups will be calculated for changes in pain, severity of digital triggering, and changes in physical function as measured through the QuickDASH.

The principal investigator of this study will be responsible for the analytical / statistical tasks.

Data Collection/ Assessment Instruments:

Master List: The Master List is a participant data sheet for all nine participants which permits the correlation of each of the nine participants with their subject ID, medical record number, and telephone number. The principal investigator will be the only individual with access to the Master List. The Master List was developed specifically for this study. The master list will be kept separate from the outcome data.

Orthotic Daily Log: A daily log to be completed by the participant of their orthotic schedule wearing compliance as well as their comfort level and functional use of their hand while wearing your orthotic. The Orthotic Daily Log was developed specifically for this study.

Home Exercise Program (HEP) Daily Log: A daily log completed by the participant of their home exercise program compliance. The HEP Daily Log was developed specifically for this study.

OCTH Project Data Collection Sheet: Participant data collection sheet for all nine participants, which will be identified only by subject ID#, permits documentation of orthotic type, gender, age (recorded as ">89" if >90 yo), trigger grade, pain, wearing schedule, and QuickDash Score. The OCTH Project Data Collection Sheet was developed specifically for this study.

Quick Dash: An eleven-item outcome measure survey of the participants symptoms and ability to perform activities completed by the participant at the time of their initial evaluation and then again at the time of their discharge from therapy to permit a pre-intervention to post-intervention assessment. The QuickDash has been validated and is commonly used for research purposes (Beaton et al., 2005).

Data Collection Resources:

All participant data collected will be performed by the principal investigator who will also be the treating therapist providing direct patient care for the participants of the study.

Data Sources:

Review of Sharp HealthCare electronic and paper medical records, physician office records, laboratory test results, diagnostic test results, radiographic imaging studies including radiology reports and radiographic images.

Privacy of Subjects:

Subjects will be recruited from the principal investigators patient population as they become available through referral for therapy and will be contacted while in the outpatient rehabilitation clinic at Sharp Chula Vista Medical Center where the research study will be conducted and the participants will be attending therapy.

A medical records review will be performed by the investigator who will also be the potential participants treating therapist. A Waiver of Authorization will be requested as the investigator will need to review the medical records prior to meeting the potential participants in order to determine if basic eligibility criteria are met. The medical records review will include Sharp HealthCare paper and electronic medical records, and physician office records. Data collected will include the names for the subjects, elements of dates directly related to the subject, medical record numbers, and the subject's medical information.

During the initial evaluation and follow-up treatment sessions information will be obtained from the subject to evaluate, assess, treat and monitor the progress of their triggering finger(s). The subject will be evaluated and treated in an open gym area where other patients will be receiving therapy, or the subject may be provided with treatment in a private room if preferred by the subject. Only the subject's upper extremities need to be exposed for the evaluation and treatment of their triggering finger(s).

Confidentiality of Data and Storage:

Each subject will be provided with a coded, sequentially numbered subject ID to maintain the confidentiality of identifiable subject information.

The subjects' identity will be kept on a Master List and will remain separate from their data. The Master List will be maintained by John Avery who is the principal investigator. The master list will remain physically locked in a secure metal cabinet located at the research site that only the principal investigator, who will also be the treating therapist, will have access to.

Upon completion of the study, all of the participants' identifiers will be destroyed which is anticipated to be 06/01/2020.

Subjects will be identified on research-related forms as follows: Master List: Subject ID, Name, MRN; HEP and Orthotic Daily Log: Subject ID only; OCTH Project Data Collection Sheet: Subject ID, Gender, Age (">89" if >90 yo).

The subject's names, social security number, medical record number, Sharp financial identification number (FIN), and any identifier (other than subjects' study identification number) will not be sent off site. This data will not be used for any other purpose, other than that for which the subjects will be consented.

Benefits to Individual Subjects:

Benefits to the subjects as a direct result of participating in the study include a more intensive monitoring of their progress and compliance with their orthotic wear and home exercise program.

Potential Benefits (Value) to Society:

This case series will provide feasibility data in preparation for a randomized controlled study of this topic in the future. Practitioners can use the information obtained through this case series as a platform for further inquiry regarding the efficacy of various wearing schedules.

Risk Category: Minimal

Potential Risks:

All risks to the participants are no greater than what would be expected clinically for participants not participating in the study, except for a slightly increased risk of loss of confidentiality due to increased assessment associated with the study.

Potential risk includes one or more of the subjects developing a pressure wound or discomfort from wearing of the custom fabricated thermoplastic orthotic on their hand.

The risk of developing a pressure wound or discomfort is associated with pressure and shear of the orthotic against the participant's tissue and the risk increases as the amount of pressure, shear and time under pressure increases.

A subject's risk for developing discomfort or a pressure wound may increase if the subject forcefully and / or repetitively flexes their digit while wearing an orthotic on it such as during a waking activity or while sleeping.

The potential for a subject to experience a pressure wound or discomfort secondary to wearing of their digital orthotic may be greater with continuous wear relative to wearing only while awake or while sleeping due to the increased total amount of time the orthotic is donned. However, a subject's individual risk level will vary depending upon the activity the subject engages in and the duration and force applied through their digit against the thermoplastic orthotic during the activity.

The estimated probability of one or more of the subjects developing a pressure wound is low, and the estimated potential for reversibility is typically high.

Protection Against Risks:

The potential for the risk of any of the subjects experiencing a pressure wound will be minimized by each orthotic being carefully custom designed to fit the individual subjects, carefully monitoring the subjects for any complications related to orthotic wear, and educating the subjects on how to wear and care for the orthotic care and to discontinue wear of the orthotic if they develop any adverse reactions including tingling, numbness, pain, edema or redness at orthotic wear site that lasts longer than 20 minutes.

The orthotics to be issued to the subjects who elect to be in the study are standard of care for the treatment of trigger finger and will be fabricated only by the principle investigator.

The orthotics will be fabricated and issued within the hand clinic treatment area during a subject's treatment appointment.

The orthotics are fabricated from a flat piece of thermoplastic which is stored in an unlocked cabinet within the hand therapy treatment area of an open outpatient rehabilitation gym.

Fabricated orthotics for a participant will not be stored within the clinic.

The custom orthotic is not a significant risk device, because all of the following are true:

The orthotic is NOT intended as an implant that presents a potential for serious risk to the health, safety, or welfare of a subject.

The orthotic is NOT purported or represented to be for a use in supporting or sustaining human life that presents a potential for serious risk to the health, safety, or welfare of a subject.

The orthotic is NOT for a use of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health that presents a potential for serious risk to the health, safety, or welfare of a subject.

The orthotic is does NOT otherwise present a potential for serious risk to the health, safety, or welfare of a subject.

The orthitic is not a banned medical device. The custom fabricated thermoplastic digital orthotic that will be fabricated and issued by the principle investigator of this study to participants with trigger finger is a standard of care for the treatment of trigger finger and has not been banned.

The custom orthotic that will be issued to the participants will be worn externally on the triggering digit(s) and are not purported or represented to be for use in supporting or sustaining human life that presents a potential for serious risk to the health, safety, or welfare of a subject.

I do not believe that trigger finger, in and of itself, presents a potential for serious risk to the health, safety, or welfare of a subject.

I do not believe that use of the custom thermoplastic orthotic to be issued by the principle investigator this study to the subjects of this study subjects presents a serious risk to their health, safety or welfare.

Consent Process The following investigators and internal staff will obtain consent: John Avery, (PI) University of Utah John Avery, who is the principal investigator, will be only person obtaining consent / assent from the participants.

Location(s) where consent will be obtained. 752 Medical Center Court, Suite 303, Chula Vista, California, 91911

Recruitment Process:

Participants will be recruited through a convenience sampling of patients as they become available to the researcher's clinic for hand therapy, meet the study's eligibility criteria and provide informed consent to participate in the study.

Medical records review will be performed by the principal investigator who will also be the potential participants' treating therapist.

All of the participant's questions relevant to the study and necessary to facilitate rational and thoughtful decision making by the participant will be answered prior to signing the consent form.

Signed consent documentation will remain physically locked in a secure metal cabinet located at the research site that only the principal investigator / treating therapist will have access to.

Potential participants will be told that participation is completely voluntary and that participating in the study will not affect the treatment they receive for their triggering digit(s).

All of the participant's questions relevant to the study and necessary to facilitate rational and thoughtful decision making by the participant will be answered prior to signing the consent form.

Prior to obtaining consent, the prospective participants will be asked if they sufficiently understand the information provided in order to make an informed decision regarding whether or not to participate in the research.

Potential participants will be allowed approximately 30 minutes during their initial evaluation / treatment session to decide they wish to participate in the research study. After the first 30 minutes of the participants 45 minute appointment, if the potential participant meets the study criteria and agrees to participate in the study, they will then be provided with care that is unique to the study participants and needs to be performed at the time of the initial evaluation including the following: signing the consent; completing the DASH; being provided with an orthotic wearing schedule (which may be different if they do not agree to participate in the study); a home exercise program log; and an orthotic wearing log. Additional time cannot be permitted beyond the 30 minutes provided to the participants to decide if they want to participate in the study due to the need to begin treatment during the first visit to be an ethical provider and meet rules regarding service provision.

Are there any no costs to the participants from participation in research? No Participants of the study will be responsible for their costs associated with attending occupational therapy for treatment of their triggering digit(s).

All study visits are standard of care in that no subject in this study will require more visits than they would have required if they were not enrolled in this study.

No study procedures performed for this study are expected to result in additional study visits and consequent additional costs to the subject.

Is there any compensation to the participants? No Does this study involve Protected Health Information (PHI) or de-identified health information? No What method(s) of authorization that will be used: (Consent and) Authorization Document Will PHI be disclosed outside the Covered Entity? No

Background/Experience of the Investigator:

The principal investigator, John Avery, is a licensed and registered occupational therapist and certified hand therapist. He received his bachelor's degree in occupational therapy in December 1996 from San Jose State University, and is currently pursuing his post-professional doctorate in occupational therapy from the University of Utah. He has practiced as an occupational therapist since 1997, specialized in hand therapy since 1998, and worked at Sharp Chula Vista Medical Center since October 2000.

The principal investigator, John Avery, in only investigator for this study and is the author of the study protocol.

John Avery completed the following training:

1. CITI Program Good Clinical Practice Course (USFDA focus), stage 1. Completed on 7/29/18. Expiration date is 7/28/21.
2. CITI Program Human Research, Group 1, Biomedical Research Investigators and Key Personnel, Basic course.

   Completed 7/29/18. Expiration date is 7/28/21.
3. HIPPA for clinicians, completed annually

ELIGIBILITY:
Inclusion Criteria:

1. referred to hand therapy with single digit triggering of left and / or right hand.
2. agreement to participate in the study and receive an orthotic as part of the treatment of digital triggering.

If after four months of utilizing the previously stated criteria all nine participants have not been able to be recruited, the criteria will be broadened. The inclusion criteria will be broadened to include:

(1) referred for hand therapy with one or more digits triggering.

Exclusion Criteria:

1. a triggering digit that presents with Froimson's (1999) grade III or IV of severity (Table 1).
2. triggering of the affected digit for greater than 6 months.
3. more than one triggering digit per hand.
4. a triggering thumb.
5. have received a corticosteroid injection in the triggering digit within the past 2 years.
6. do not speak English.
7. a diagnosed cognitive deficit that impairs their ability to follow the protocol of the study and provide informed consent to participate in the study.
8. less than 18 years of age.

If after four months of utilizing the previously stated criteria all nine participants have not been able to be recruited, the criteria will be broadened. The exclusion criteria will be broadened to include:

(1) a triggering digit that is locked in flexion and unable to be passively unlocked; Froimson's (1999) grade IV.

Table 1 Froimson's (1999) grading of digital triggering severity

Grade I: Pain associated with pre-triggering. Tenderness to palpation over the first annular pulley. Reported history of digital triggering, although not reproducible during clinical examination.

Grade II: Digital triggering occurs, although, digit can be unlocked with active extension.

Grade III: Digital triggering occurs and passive extension is necessary to unlock the digit, or active flexion is unable to be performed at the digit.

Grade IV: Digital triggering of the interphalangeal joint is unable to be unlocked with active or passive movement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
The amount of time in weeks it took to enroll the nine participants. | up to 8 months (anticipated)
  To assist with determining the feasibility of the study, the rate at which participants become available for the study will be measured, analyzed and reported through descriptive statistics.
The participants' functional use of their hand and comfort while wearing their orthotic. | up to 8 months (anticipated)
  To permit measuring the comfort of the orthotic and the participants functional use of their hand while wearing the orthotic, the participants will be asked to complete a daily log.
  The participants' functional use of their hand and comfort while wearing their orthotic will be included in the data analysis and reported through descriptive statistics to assist with determining the feasibility of the study,
The participants' percentage compliance with their prescribed wearing schedules. | up to 8 months (anticipated)
  To permit measuring the participants' compliance with their prescribed HEP performance schedule, the participants will be asked to complete a daily check-box log.
  To assist with determining the feasibility of the study, the participants' percentage compliance with their prescribed wearing schedules will be analyzed and reported through descriptive statistics.
The participants' percentage compliance with their HEP performance schedule | up to 8 months (anticipated)
  To permit measuring the participants' compliance with their prescribed HEP performance schedule, the participants will be asked to complete a daily check-box log.
  To assist with determining the feasibility of the study, The participants' percentage compliance with their HEP performance schedule will be analyzed and reported through descriptive statistics.

SECONDARY OUTCOMES:
Participant outcome measure: Participant pain levels | up to 8 months (anticipated)
  NPRS will be used to measure participant pain levels. The NPRS utilized ranges from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable (Young, Cleland, Michener, & Brown, 2010). The NRPS has been shown to be a reliable and valid measure of pain (Ferreira-Valente, Pais-Ribeiro & Jensen, 2011; Jensen, Karoly & Braver, 1986; Young et al., 2010).
Participant outcome measure: Participant trigger finger severity | up to 8 months (anticipated)
  Froimson's (1999) scale will be used to measure triggering across four grades of severity (Table 1). Yang et al. (2014) demonstrated that the severity of Froimson's (1999) grade III and IV, as well as grade II when insufficiently responsive to three months of conservative treatment, was correlated with the grading of affected pathological full thickness A-1 pulley tissue samples.
Participant outcome measure: QuickDASH for the measurement of upper extremity symptoms and disability | up to 8 months (anticipated)
  QuickDASH (Disabilities of the Arm, Shoulder and Hand Outcome Measure): An eleven-item outcome measure survey of the participants symptoms and ability to perform activities completed by participant at the time of their initial evaluation and then again at the time of their discharge from therapy.
  QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high-performance sport/music or work modules (4 items, scored 1-5).
  Disability/Symptom section: Assigned values for all completed responses are summed and averaged, producing a score out of five. This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. A higher score indicates greater disability. = sum of n responses - 1 x 25, n where n is equal to the number of completed responses.
  Optional modules: For each module add up the assigned values for each response and divide by four; subtract one and multiply by 25 to obtain a score out of 100.

CONTACTS AND LOCATIONS:
Overall Officials: John C Avery, BS, Principal Investigator — Sharp Chula Vista Medical Center
Locations (1):
- Sharp Chula Vista Medical Center Outpatient Rehabilitation Department, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams JE, Habbu R. Tendinopathies of the Hand and Wrist. J Am Acad Orthop Surg. 2015 Dec;23(12):741-50. doi: 10.5435/JAAOS-D-14-00216. Epub 2015 Oct 28. PMID 26510626
- [Background] Akhtar S, Bradley MJ, Quinton DN, Burke FD. Management and referral for trigger finger/thumb. BMJ. 2005 Jul 2;331(7507):30-3. doi: 10.1136/bmj.331.7507.30. No abstract available. PMID 15994689
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Colbourn J, Heath N, Manary S, Pacifico D. Effectiveness of splinting for the treatment of trigger finger. J Hand Ther. 2008 Oct-Dec;21(4):336-43. doi: 10.1197/j.jht.2008.05.001. Epub 2008 Aug 22. PMID 19006759
- [Background] Evans, R., Hunter, J., & Burkhalter, W. (1988). Conservative management of the trigger finger: A new approach. Journal of Hand Therapy, 59-68.
- [Background] Drijkoningen T, van Berckel M, Becker SJE, Ring DC, Mudgal CS. Night Splinting for Idiopathic Trigger Digits. Hand (N Y). 2018 Sep;13(5):558-562. doi: 10.1177/1558944717725374. Epub 2017 Aug 20. PMID 28825334
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Froimson, A. (1999). Tenosynovitis and tennis elbow. In: Green, D.P., et al. (eds.), Green's Operative Hand Surgery, wyd. 4. Churchill Livingstone.
- [Background] Huisstede BM, van Middelkoop M, Randsdorp MS, Glerum S, Koes BW. Effectiveness of interventions of specific complaints of the arm, neck, and/or shoulder: 3 musculoskeletal disorders of the hand. An update. Arch Phys Med Rehabil. 2010 Feb;91(2):298-314. doi: 10.1016/j.apmr.2009.09.023. PMID 20159137
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Kim SJ, Lee CH, Choi WS, Lee BG, Kim JH, Lee KH. The thickness of the A2 pulley and the flexor tendon are related to the severity of trigger finger: results of a prospective study using high-resolution ultrasonography. J Hand Surg Eur Vol. 2016 Feb;41(2):204-11. doi: 10.1177/1753193415615076. Epub 2015 Nov 14. PMID 26568540
- [Background] Lieberman D, Scheer J. AOTA's Evidence-Based Literature Review Project: an overview. Am J Occup Ther. 2002 May-Jun;56(3):344-9. doi: 10.5014/ajot.56.3.344. No abstract available. PMID 12058525
- [Background] Makkouk AH, Oetgen ME, Swigart CR, Dodds SD. Trigger finger: etiology, evaluation, and treatment. Curr Rev Musculoskelet Med. 2008 Jun;1(2):92-6. doi: 10.1007/s12178-007-9012-1. PMID 19468879
- [Background] Patel MR, Bassini L. Trigger fingers and thumb: when to splint, inject, or operate. J Hand Surg Am. 1992 Jan;17(1):110-3. doi: 10.1016/0363-5023(92)90124-8. PMID 1538090
- [Background] Rodgers JA, McCarthy JA, Tiedeman JJ. Functional distal interphalangeal joint splinting for trigger finger in laborers: a review and cadaver investigation. Orthopedics. 1998 Mar;21(3):305-9; discussion 309-10. doi: 10.3928/0147-7447-19980301-13. PMID 9547815
- [Background] Ryzewicz M, Wolf JM. Trigger digits: principles, management, and complications. J Hand Surg Am. 2006 Jan;31(1):135-46. doi: 10.1016/j.jhsa.2005.10.013. PMID 16443118
- [Background] Sato J, Ishii Y, Noguchi H, Takeda M. Sonographic appearance of the flexor tendon, volar plate, and A1 pulley with respect to the severity of trigger finger. J Hand Surg Am. 2012 Oct;37(10):2012-20. doi: 10.1016/j.jhsa.2012.06.027. Epub 2012 Aug 31. PMID 22939830
- [Background] Tarbhai K, Hannah S, von Schroeder HP. Trigger finger treatment: a comparison of 2 splint designs. J Hand Surg Am. 2012 Feb;37(2):243-9, 249.e1. doi: 10.1016/j.jhsa.2011.10.038. Epub 2011 Dec 20. PMID 22189188
- [Background] Valdes K. A retrospective review to determine the long-term efficacy of orthotic devices for trigger finger. J Hand Ther. 2012 Jan-Mar;25(1):89-95; quiz 96. doi: 10.1016/j.jht.2011.09.005. PMID 22265444
- [Background] Yang TH, Chen HC, Liu YC, Shih HH, Kuo LC, Cha S, Yang HB, Yang DS, Jou IM, Sun YN, Su FC. Clinical and pathological correlates of severity classifications in trigger fingers based on computer-aided image analysis. Biomed Eng Online. 2014 Jul 23;13:100. doi: 10.1186/1475-925X-13-100. PMID 25055721
- [Background] Young IA, Cleland JA, Michener LA, Brown C. Reliability, construct validity, and responsiveness of the neck disability index, patient-specific functional scale, and numeric pain rating scale in patients with cervical radiculopathy. Am J Phys Med Rehabil. 2010 Oct;89(10):831-9. doi: 10.1097/PHM.0b013e3181ec98e6. PMID 20657263